CLINICAL TRIAL: NCT03889795
Title: Phase IB Trial of Metformin, Digoxin, Simvastatin in Subjects With Advanced Pancreatic Cancer and Other Advanced Solid Tumors
Brief Title: Phase IB Metformin, Digoxin, Simvastatin in Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Danae Hamouda, MD (Other)
Responsible Party: Sponsor-Investigator, Danae Hamouda, MD, Principal Investigator and Medical Director, University of Toledo
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Advanced Pancreatic Cancer; Advanced Solid Tumor
Keywords: Pancreatic; Solid Tumor; Advanced Pancreatic Cancer; Dose Escalation; Maximum Tolerated Dose
MeSH Terms: interventions — Metformin; Simvastatin; Digoxin

STUDY DESIGN:
Intervention Model Description: 3 Subjects per Cohort + 3 additional subjects in Expansion Cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose Escalation (Experimental): C3 (Metformin, Simvastatin and Digoxin) will be dosed each day of a 28 calendar day cycle. The starting dose level will be increased with each cohort. There are 3 cohorts. Upon reaching maximum tolerated dose, an expansion cohort will be opened. Cohort 1 - Metformin 850mg po/day, Simvastatin 5mg po/day, Digoxin 0.0625 mg po/day. Cohort 2 - Metformin 850 mg po/day for two weeks and 1,700 mg po/day for next two weeks, Simvastatin 20 mg po/day, Digoxin 0.25 mg po/day. Cohort 3 - Metformin 850 mg po/day for two weeks and 1,700 mg po/day for next two weeks, Simvastatin 40 mg po/day, Digoxin 0.25 mg po/day for two weeks, 0.375 mg po/day for the next two weeks for cycle 1. Subjects will receive 0.50 mg po/day in Cohort 3, Cycle 2 and beyond. Metformin to be taken at Breakfast and Dinner time (as applicable), Simvastatin at Bed time and Digoxin once daily.
  Interventions: Drug: Metformin; Drug: Simvastatin; Drug: Digoxin

INTERVENTIONS:
Drug: Metformin — Metformin oral pill will be taken daily at breakfast (cohort 1) and breakfast and dinner (cohort 2 and 3).
  Other Names: Glucophage
Drug: Simvastatin — Simvastatin oral pill will be taken daily in the evening.
  Other Names: Zocor
Drug: Digoxin — Digoxin oral pill will be taken once daily.
  Other Names: Digitalis

SUMMARY:
This is a single-center trial in subjects with pancreatic cancer and other advanced solid tumors. It is an open-label, single arm dose escalation Phase IB trial with subjects accrued in a 3 subject dose escalation cohort. Subjects with treated advanced solid tumors, and showing disease progression on established standard therapy, will be enrolled in this trial.

DETAILED DESCRIPTION:
This is a single-center trial in subjects with pancreatic cancer and other advanced solid tumors. It is an open-label, single arm dose escalation Phase IB trial with subjects accrued in a 3 subject dose escalation cohort. Subjects with treated advanced solid tumors, and showing disease progression on established standard therapy, will be enrolled in this trial.

C3 (Simvastatin + Digoxin + Metformin) will be given as three oral pills within recommended package insert safe levels. Subjects will be accrued in 3-subject dose escalation cohorts. 3 additional subjects will be treated at the presumptive maximum effective cohort dose/schedule for a total of 6 subjects at maximum effective level.

ELIGIBILITY:
Inclusion Criteria

1. Subject ≥18 years with histologically confirmed solid tumor.
2. Dose expansion subjects must have at least one tumor mass amenable to core needle biopsy.
3. Refractory or intolerant to established standard of care.
4. Have at least one tumor mass amenable to core needle biopsy. Adequate Archival Tissue required for patients that will take part in the dose escalation cohorts.
5. ECOG performance status (PS) = 0-2, or Karnofsky PS ≥60%, or Lansky PS ≥60%.
6. Normal organ and marrow function: absolute granulocyte count ≥1,000/mm3, absolute lymphocyte count ≥400/mm3, platelets ≥100,000/mm3, total bilirubin ≤ institutional upper normal limit, AST/ASL ≤2x institutional upper limit of normal, GFR >60 mL/min/1.73 m2 and creatinine <1.5 mg/dL.
7. Subject has recovered to CTCAE Grade 1 or better from all adverse events associated with prior therapy or surgery. Pre-existing motor or sensory neurologic pathology or symptoms must be recovered to CTCAE Grade 2 or better.
8. If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will then be required for study entry.
9. Ability to understand and the willingness to sign a written informed protocol specific consent.

Exclusion Criteria:

1. Anti-cancer chemotherapy, biologic therapy or immunotherapy within 3 weeks or radiation therapy within 2 weeks of first infusion.
2. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
3. Patients with only PET non-avid disease.
4. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months.
5. Known history of rhabdomyolysis.
6. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the Investigator.
7. Known HIV or chronic Hepatitis B or C infection.
8. Have signs and symptoms consistent with an active infection.
9. Live vaccination for the prevention of infectious disease administered <30 days prior to the start of study therapy or inactivated vaccination <14 days prior to the start of study therapy.
10. History of severe allergic, anaphylactic, or other hypersensitivity reactions to Metformin, Simvastatin, and/or Digoxin.
11. Patients diagnosed with Wolff-Parkinson-White Syndrome or electrocardiographic (ECG) pattern. Other cardiac conditions including: Previous MI with evidence of residual electrographic pattern consisted with bradycardia/heart block. Atrio-ventricular (AV) heart block (currently ongoing). History of ventricular fibrillation. Sick Sinus Syndrome or Sinus bradycardia thought to be caused by sinus node disease, unless effectively treated. Heart failure associated with preserved left ventricular ejection fraction, including constructive pericarditis, restrictive cardiomyopathy, and Amyloid heart muscle disease.
12. Women of childbearing potential who are found to be pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and/or Recommended Dose within the tested C3 dose range | Up to one year
  Occurrence of any ≥ Grade 3 toxicity encountered within the four weeks following the administration of C3, regardless of attribution

SECONDARY OUTCOMES:
Safety and Tolerability: Occurrence of treatment - emergent adverse events (TEAEs) and other abnormalities | Up to 2 years
  Occurrence of treatment - emergent adverse events (TEAEs) and occurrence of abnormalities in laboratory test values, markedly abnormal vital sign measurements, and clinically significant abnormal electrocardiograms (ECGs), including conduction abnormalities and changes in QT interval
Efficacy (Disease Response) | Up to 2 years
  Response and progression evaluated using Response Evaluation criteria in solid tumors
Assess BIRC5 levels of expression in tumor tissue | RNA and protein levels of expression at baseline and at 2 months after C3 treatment
  Blood samples for pharmacokinetic analysis of C3 will be collected at designated time points.
Assess molecular changes induced by C3 administration in the blood for biomarker sensitivity/resistance assessment | Baseline and at 2 months
  Molecular signal tumor blood (plasma) and microenvironment protein expression patterns via quantitative mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Danae Hamouda, MD, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Eleanor N. Dana Cancer Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No